CLINICAL TRIAL: NCT04435262
Title: Syncope and Implanted Loop Recorder: the Utility of Remote Monitoring and Patients Centered Setting Alarms in Real World Setting.
Brief Title: Syncope and Implanted Loop Recorder: the Utility of Remote Monitoring and Patients Centered Setting Alarms
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Vincenzo Russo, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: 181060320
Record Dates: First submitted 2020-06-10; First posted 2020-06-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Syncope; Loop Recorder; Remote Monitoring
Keywords: Syncope; Loop Recorder; Remote Monitoring
MeSH Terms: conditions — Syncope | interventions — Remote Patient Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ILR Group followed with RM: Patients with unexplained syncope underwent ILR monitoring and followed with RM
  Interventions: Other: Remote Monitoring
- ILR Group followed with in-hospital visits: Patients with unexplained syncope underwent ILR monitoring and followed with in-hospital visits

INTERVENTIONS:
Other: Remote Monitoring — Remote Monitoring Follow-up
  Groups: ILR Group followed with RM

SUMMARY:
Actually, there are few data about the effectiveness of remote monitoring (RM) and patient centered alarms setting in patients with unexplained syncope underwent implanted loop recorder (ILR) monitoring.

The aim of this study is to evaluate the time from onset of first physician's evaluation of asyntomatic ECG events lead to medical treatment in ordinary clinical practice for syncope patients with ILR patients and compare it between patients followed with RM or conventionally with annual in-hospital visits.

ELIGIBILITY:
Inclusion Criteria

* Patients with unexplained syncope underwent ICM implantation according to current gudelines.

Exclusion Criteria

* Patients do not provied signing Patient Informed Consent Form

Min Age: 14 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population included all patients with unexplained syncope underwent ICM implantation according to current gudelines and followed by conventionally or RM according to the hospital's clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-05-10 (Actual); Primary Completion 2022-03-16 (Estimated); Study Completion 2024-03-16 (Estimated)

PRIMARY OUTCOMES:
Time to medical treatment | through study completion, an average of 1 year
  Time from onset of first physician's evaluation of asyntomatic ECG events lead to medical treatment in ordinary clinical practice for syncope patients with ILR patients and compare it between patients followed with RM or conventionally with annual in-hospital visits.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Campania "Luigi Vanvitelli", Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided